CLINICAL TRIAL: NCT06790225
Title: Glucose-dependent INsulinotropic Polypeptide: Effect on Bone Remodelling and Cell Activity (GINEBRA)
Acronym: GINEBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 25/2685
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Bone Disease, Metabolic; Diabetes Mellitus, Type 2; Obesity and Obesity-related Medical Conditions
Keywords: GIP; CTX; P1NP; Glucose-dependent insulinotropic polypeptide; Bone remodelling
MeSH Terms: conditions — Bone Diseases, Metabolic; Diabetes Mellitus, Type 2; Obesity | interventions — Incretins

STUDY DESIGN:
Intervention Model Description: Participants are randomized to recive either intermittent ( 8 hours a day) or continious (24 hours a day) GIP infusion for three days. The effect of GIP will be measured by bone markers in blood samples, as well as in vitro activity and genetic alterations of bone cells using bone marrow aspirates and bone marrow biopsies. Each participant will recive both administrations using a crossover design with 14-28 days washout period inbetween.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent then continious (Experimental): The participants that recive the intermittent administration first, followed by the continious
  Interventions: Other: Glucose-dependent Insulinotropic Polypeptide (GIP)
- Continious then intermittent (Experimental): The participants that recives the continious administration first, follwoed by the intermittent
  Interventions: Other: Glucose-dependent Insulinotropic Polypeptide (GIP)

INTERVENTIONS:
Other: Glucose-dependent Insulinotropic Polypeptide (GIP) — Recombinant human GIP (1-42)

SUMMARY:
Glucose-dependent insulinotropic polypeptide (GIP) is released by the intestines in response to food intake and increases insulin secretion. Although short-term (< 3 hours) stimulation with GIP decreases bone resorption in humans, the effect may vanish following continuous administration within 24 hours, at least in patients with type 1 diabetes. Whether the anti-resorptive effect of GIP can be maintained if the hormone is non-continuously administrated is unclear. As the first GIP receptor (GIPR) agonist, tirzepatide was recently approved for the treatment of obesity and type 2 diabetes in the USA and type 2 diabetes alone in the EU, there is a need to establish knowledge about the long-term effects of GIP on bone health, including if different exposure times to GIP have different skeletal effects.

This project will investigate whether GIP maintains its anti-resorptive potential if given as intermittent compared to continuous infusion in healthy men and women aged 18-40 years. Administration cycles involve intermittent (8 hours daily) and continuous (24 hours daily) injection of GIP for three days each. The effect of GIP will be measured by bone markers in blood samples, as well as in vitro activity and genetic alterations of bone cells (osteoclasts and osteoblasts) using bone marrow aspirates and bone marrow biopsies. Each participant will receive both administration cycles using a crossover design with a 14-28 days washout period between administrations of GIP.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pre-diabetes or diabetes (HbA1c >42mmol/mol)
* BMI >28
* fractures with < 6months
* comorbidities/treatments that may influence bone metabolism or procedures - -- pregnancy
* inability to provide informed concent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of CTX | During a three day period. With 14-28 days of washout between the two administration methods
  Serum levels of CTX (bone resorption marker) will be measured prior to, during, and at after the intervention, with both administration methods (continious and intermittent)

SECONDARY OUTCOMES:
Serum levels of osteocalcin and P1NP | During a three day period. With 14-28 days of washout between the two administration methods
  Serum levels of osteocalcin and P1NP (bone formation markers) will be measured prior to, during, and at after the intervention, with both administration methods (continious and intermittent)
Serum levels of GIP | During a three day period. With 14-28 days of washout between the two administration methods
  Serum levels of GIP will be measured prior to, during, and at after the intervention, with both administration methods (continious and intermittent)

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Southern Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared following GDPR and local data mangament regulation. However data(anonymous) and results will be published once the study is completed.